CLINICAL TRIAL: NCT03640988
Title: A Post-market Pilot Study to Evaluate the Effects of High Energy Acoustic Shock Wave Therapy on Local Skin Perfusion and Healing of Diabetic Foot Ulcers
Brief Title: The Effects of High Energy Acoustic Shock Wave Therapy on Local Skin Perfusion and DFUs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Mfr of product identified in protocol to measure perfusion after treatment with sponsor device withdrew support from the study. Sponsor decided to cancel the investigation due to lack of adequate replacement.
Sponsor: SANUWAVE, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAN18-DERM02
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Pulsed acoustic wave on-label application on acute and chronic defects of the skin and subcutaneous soft tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- dermaPACE (Experimental): Non-sterile, single, Benchtop System that is comprised of a dermaPACE Control Console, PACE Applicator and foot pedal. The PACE applicator uses shockwave technology on acute and chronic defects.
  Interventions: Device: dermaPACE

INTERVENTIONS:
Device: dermaPACE — Shockwave application

SUMMARY:
This is an observational, single-arm, on-label study. This clinical study will be conducted at up to 2 sites with a total of 10 subjects per site. All subjects will receive standard of care treatment which includes DFU treatments with the dermaPACE device.

DETAILED DESCRIPTION:
The dermaPACE system will be used according to label along with standard of care. perfusion will be measured using TcPO2 methods and also using cleared hyperspectral imaging equipment. The intent of the study is to observe/measure oxygen saturation levels in the area of the treated wound before initiation of dermaPACE treatment, during the treatment period, and two weeks post treatment period

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female ≥22 years of age at Visit 1;
2. Wagnergrade 1 or 2 DFU;
3. In the leg with the target ulcer has an ABI > 0.70 and < 1.20 OR if the ABI is >1.20 has a toe pressure >50 mmHg at Visit 1
4. Has only one diabetic foot ulcer that is located on the plantar surface of the forefoot that has persisted a minimum of 30 days prior to the first visit.
5. Has Type I or Type II Diabetes Mellitus;
6. HbA1c < 12% at Visit 1;
7. Patient is willing to comply with all study requirements and treatment visits.
8. Patient is willing to comply with off-loading directions.
9. Patient is willing to comply with offloading instructions

Exclusion Criteria:

* Potential subjects who meet any of the following criteria will be excluded from participating in the study.

A subject who:

1. Is female and is currently pregnant or plans to become pregnant during the study;=, or is a female who is nursing aor actively lactating;
2. Known or suspected systemic infection;
3. Enrolled in another investigational study;
4. Has received growth factor therapy (e.g., autologous platelet-rich plasma, stem cell therapy, becaplermin, cell therapy, dermal substitute, amniotic tissue, extracellular matrix) within 30 days of study enrollment;
5. Subject is currently receiving or has received radiation or chemotherapy within 3 months of study enrollment;
6. Unable to tolerate offloading footwear or total contact casting (TCC);
7. Has active cellulitis either at the site of, or in the surrounding area of, the target ulcer at Visit 1 or 2;
8. Has active Charcot foot at Visit 1 or 2;
9. Has osteomyelitis in the foot or ankle on which the target ulcer is located at Visit 1 or 2

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-01-03 (Actual)

PRIMARY OUTCOMES:
Skin perfusion, effect on oxygenation level, by visit | 10 weeks
  Measurement of changes in oxygenation levels in superficial tissue before and after treatment with dermaPACE System.

SECONDARY OUTCOMES:
Wound healing, effect on wound area, by visit | 10 weeks
  Measurement of changes in wound area at each visit
Wound healing, effect on wound closure, by visit | 10 weeks
  Measurement of the rate of wound closure at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Mark Granick, MD FACS, Principal Investigator — University Hospital/Rutgers University
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No